CLINICAL TRIAL: NCT02942472
Title: Position Of The Tip Of The Inner Catheter And Air Bubbles As Predictors Of Pregnancy During ICSI Cycles:Prospective Observational Study
Brief Title: Position Of The Tip Of The Inner Catheter And Air Bubbles As Predictors Of Pregnancy During ICSI Cycles
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, AMR HELMY YEHIA, Associate Professor, Ain Shams Maternity Hospital
Other Study IDs: MOHEgypt
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Pregnancy
Keywords: clinical pregnancy rate after embryo transfer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Position of the tip of the inner catheter and air bubbles detection (at time,5min 10min)during embryo transfer influence the pregnancy rate in ICSI cycles .

DETAILED DESCRIPTION:
The aim of this study is to assess the relationship between the position of the tip of the inner catheter, the position of the air bubbles (at time , 5 min ,10 min )after embryo transfer and pregnancy rate outcome in ICSI cycles. Most IVF teams consider not touching the endometrium and the uterine fundus with replacement of the embryos in the lumen of the endometrial cavity the most important factors for successful embryo transfer, it is highly recommended to use agents that can facilitate a smooth embryo transfer and reduce unintended stimulation of the fundus, for example the application of soft-tipped catheters, which can improve pregnancy rate.

The advantage of using the air and liquid content for catheter loading is to prevent the embryo from adhering to the wall of the catheter at the time of injection.The presence of two air bubbles on both sides of the medium that contains the embryo prevents the transfer of the embryo within the catheter and beside, in the transfer under ultrasonographic guidance, the air bubbles are often considered a marker for the embryo's position in the uterus.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30 kg/ m2.
* Between 20 and 35years old.
* FSH levels on cycle day 3 of <12 mIU/mL.
* Both ovaries present deprived of morphological abnormalities and adequately visualized in Transvaginal ultrasound.
* Grade one or two embryo quality.

Exclusion Criteria:

* Hydrosalpinx.
* Intrauterine lesion.
* Patients undergoing ET after cryopreservation.
* Blood present on the catheter during the transfer procedure.
* A difficult transfer or with a suspicion of touching the fundus.
* Endometrial thickness less than 8mm.
* Known allergic reaction against one of the ingredient of the medications used during the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: prospective observational study
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | one and half year

IPD SHARING:
Plan to Share IPD: Yes